CLINICAL TRIAL: NCT02418676
Title: Insulin Complexation With Hydroxypropyl-beta-cyclodextrin: Spectroscopic Evaluation of Molecular Inclusion and Use of the Complex in Gel for Healing of Pressure Ulcers
Brief Title: Insulin Complexation With Hydroxypropyl-beta-cyclodextrin: Use of the Complex in Gel for Healing of Pressure Ulcers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: State University of Maringá (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Financiadora de Estudos e Projetos (Other); Fundação Araucária (Other)
Responsible Party: Principal Investigator, Graciette Matioli, Professor, State University of Maringá
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UEM-LaBE-01; 0069.0.093.000-11 (Other Grant/Funding Number: Ethics in Research Involving Human Subjects (SISNEP)); 035/2012 (Other Grant/Funding Number: Ethics in Research Involving Human Subjects (COPEP-UEM)); 072/2013 (Other Grant/Funding Number: HUM-COREA)
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: Pressure Ulcer; Wound
Keywords: Human insulin; Hydroxypropyl-beta-cyclodextrin; Pressure Ulcer; Wound Healing; Gel
MeSH Terms: conditions — Pressure Ulcer; Wounds and Injuries; Insulin Resistance | interventions — Gels; Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gel with HPβCD-I complex (Experimental): A quantity of 5 grams of gel with hydroxypropyl-beta-cyclodextrin complexed with insulin (HPβCD-I) was placed on the pressure ulcer, previously cleaned with saline, and covered with sterile gauze and a transparent film.
  Interventions: Drug: Gel with HPβCD-I complex
- Gel with insulin (Active Comparator): A quantity of 5 grams of gel with insulin was placed on the pressure ulcer, previously cleaned with saline, and covered with sterile gauze and a transparent film.
  Interventions: Drug: Gel with insulin
- Control gel (Placebo Comparator): A quantity of 5 grams of gel without active was placed on the pressure ulcer, previously cleaned with saline, and covered with sterile gauze and a transparent film.
  Interventions: Drug: Control gel

INTERVENTIONS:
Drug: Gel with HPβCD-I complex — Initially, the pressure ulcer was cleaned with saline. With the aid of a paper ruler, the ulcer was measured and photographed, as the ruler included the date and the initials of the patient. After measuring, a quantity of 5 grams of gel with hydroxypropyl-beta-cyclodextrin complexed with insulin (HPβCD-I) was placed on the pressure ulcer and covered with sterile gauze and a transparent film.
  The curative was changed once a day during the treatment period, unless there was leakage of fluid, contamination, or signs of infection. Every three days the pressure ulcers of all patients were measured and photographed again, resulting in a total of six measurements per patient. The photos of pressure ulcers were evaluated for measurement of pressure ulcers and any kind of irritation.
  Arms: Gel with HPβCD-I complex
Drug: Gel with insulin — Initially, the pressure ulcer was cleaned with saline. With the aid of a paper ruler, the ulcer was measured and photographed, as the ruler included the date and the initials of the patient. After measuring, a quantity of 5 grams of gel with insulin was placed on the pressure ulcer and covered with sterile gauze and a transparent film.
  The curative was changed once a day during the treatment period, unless there was leakage of fluid, contamination, or signs of infection. Every three days the pressure ulcers of all patients were measured and photographed again, resulting in a total of six measurements per patient. The photos of pressure ulcers were evaluated for measurement of pressure ulcers and any kind of irritation.
  Arms: Gel with insulin
Drug: Control gel — Initially, the pressure ulcer was cleaned with saline. With the aid of a paper ruler, the ulcer was measured and photographed, as the ruler included the date and the initials of the patient. After measuring, a quantity of 5 grams of control gel was placed on the pressure ulcer and covered with sterile gauze and a transparent film.
  The curative was changed once a day during the treatment period, unless there was leakage of fluid, contamination, or signs of infection. Every three days the pressure ulcers of all patients were measured and photographed again, resulting in a total of six measurements per patient. The photos of pressure ulcers were evaluated for measurement of pressure ulcers and any kind of irritation.
  Arms: Control gel

SUMMARY:
The coprecipitation method was used to prepare hydroxypropyl-beta-cyclodextrin complexed with insulin (HPβCD-I) by mixing insulin with hydroxypropyl-beta-cyclodextrin (HPβCD) in the molar ratio of 1:5 with the addition of 10 mL of purified water for every 100 mg of the complex. After complete dissolution of the material, the mixture was stirred for 30 min at room temperature (25°C), then left to rest for 60 min and lyophilized.

The gel was prepared by dispersing the Carbopol 940® polymer in a known amount of purified water. Under mild heating the methylparaben (0.02%, w/v), propylparaben (0.01%, w/v) and propylene glycol were dissolved and incorporated in the dispersion of Carbopol 940® and left to rest for a period of 12h. After this time, the prepared gel was stirred and pH corrected to a range of 5.0 to 7.0 with triethanolamine. A set amount of insulin and the HPβCD-I complex were incorporated into the control gel for the preparation of other formulations.

A randomized, double-blind, prospective clinical trial was conducted from March 2013 to April 2014 at the Hospital Universitário Regional de Maringá (HUM), Paraná, Brazil, in order to determine the safety and efficacy of gel in patients hospitalized in the Intensive Care Unit.

Hyperglycemic volunteers and those with pressure ulcers other than grade II were excluded from the study. Grade II pressure ulcers were selected as they are a superficial lesion, with little tissue loss, and allow easy visualization of healing.

A letter of free and informed consent was obtained. The study was conducted with each patient for a period of 15 days.

The volunteers were divided equally into three groups A, B and C, with each group being formed by five volunteers (n=5). Group A was randomly selected for treatment with gel with HPβCD-I complex, group B for treatment with gel with insulin, and group C with the control gel.

Blood glucose tests were performed in order to assess whether the insulin complexed or otherwise with HPβCD could cause an increase in the rate of insulin in the blood in patients, leading to hypoglycemia.

An identical standardized procedure for gel placement was used for all patients. Initially, the pressure ulcer was cleaned with saline. With the aid of a paper ruler, the ulcer was measured and photographed, as the ruler included the date and the initials of the patient. After measuring, a quantity of 5 grams of gel was placed on the pressure ulcer and covered with sterile gauze and a transparent film.

The curative was changed once a day during the treatment period, unless there was leakage of fluid, contamination, or signs of infection. Every three days the pressure ulcers of all patients were measured and photographed again, resulting in a total of six measurements per patient. The photos of pressure ulcers were evaluated for measurement of pressure ulcers and any kind of irritation. At the end of this stage, the properly gathered study data was interpreted using the analysis software Mobile Wound Analyzer® (MOWA).

Data was evaluated by variance analysis (ANOVA), and means were compared with the Tukey test (p < 0.05) using the software Statistica 8.0/2008 (Stat Soft Inc., Tulsa, USA).

Mixed model repeated measures methodology with some covariance structures was adopted for statistical analysis of the clinical trial (p < 0.05). The Statistical Analysis System (SAS) for Windows, version 9.3 (SAS Inc., Chicago, IL) program was used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Brazilian,
* bedridden,
* of both genders,
* aged between 45 and 75 years old, and
* diabetic or not.

Exclusion Criteria:

* hyperglycemic volunteers, and
* those with pressure ulcers other than grade II.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graciette Matioli, Doctor, Study Director — State University of Maringá

REFERENCES:
- [Background] Zhang L, Zhu W, Song L, Wang Y, Jiang H, Xian S, Ren Y. Effects of hydroxylpropyl-beta-cyclodextrin on in vitro insulin stability. Int J Mol Sci. 2009 May 6;10(5):2031-2040. doi: 10.3390/ijms10052031. PMID 19564937
- [Background] Chaudhary H, Rohilla A, Rathee P, Kumar V. Optimization and formulation design of carbopol loaded Piroxicam gel using novel penetration enhancers. Int J Biol Macromol. 2013 Apr;55:246-53. doi: 10.1016/j.ijbiomac.2013.01.015. Epub 2013 Jan 31. PMID 23376559
- [Background] Siritientong T, Angspatt A, Ratanavaraporn J, Aramwit P. Clinical potential of a silk sericin-releasing bioactive wound dressing for the treatment of split-thickness skin graft donor sites. Pharm Res. 2014 Jan;31(1):104-16. doi: 10.1007/s11095-013-1136-y. Epub 2013 Jul 31. PMID 23900888

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized, double-blind, prospective clinical trial was conducted from March 2013 to April 2014 at the Hospital Universitário Regional de Maringá (HUM), Paraná, Brazil, in order to determine the safety and efficacy of gel in patients hospitalized in the Intensive Care Unit.
Pre-assignment Details: The volunteers were Brazilian, bedridden, both genders, between 45 and 75 years old and diabetic or not. Hyperglycemic volunteers and those with pressure ulcers other than grade II were excluded from the study. Grade II pressure ulcers were selected as they are a superficial lesion, with little tissue loss, and allow easy visualization of healing.
Groups:
- Gel With HPβCD-I Complex: A quantity of 5 grams of gel with hydroxypropyl-beta-cyclodextrin complexed with insulin (HPβCD-I) was placed on the pressure ulcer, previously cleaned with saline, and covered with sterile gauze and a transparent film.
  Gel with HPβCD-I complex: Initially, the pressure ulcer was cleaned with saline. With the aid of a paper ruler, the ulcer was measured and photographed, as the ruler included the date and the initials of the patient. After measuring, a quantity of 5 grams of gel with HPβCD-I complex was placed on the pressure ulcer and covered with sterile gauze and a transparent film.
  The curative was changed once a day during the treatment period, unless there was leakage of fluid, contamination, or signs of infection. Every three days the pressure ulcers of all patients were measured and photographed again, resulting in a total of six measurements per patient. The photos of pressure ulcers were evaluated for measurement of pressure ulcers and any kind of irritation.
- Gel With Insulin: A quantity of 5 grams of gel with insulin was placed on the pressure ulcer, previously cleaned with saline, and covered with sterile gauze and a transparent film.
  Gel with insulin: Initially, the pressure ulcer was cleaned with saline. With the aid of a paper ruler, the ulcer was measured and photographed, as the ruler included the date and the initials of the patient. After measuring, a quantity of 5 grams of gel with insulin was placed on the pressure ulcer and covered with sterile gauze and a transparent film.
  The curative was changed once a day during the treatment period, unless there was leakage of fluid, contamination, or signs of infection. Every three days the pressure ulcers of all patients were measured and photographed again, resulting in a total of six measurements per patient. The photos of pressure ulcers were evaluated for measurement of pressure ulcers and any kind of irritation.
- Control Gel: A quantity of 5 grams of gel without active was placed on the pressure ulcer, previously cleaned with saline, and covered with sterile gauze and a transparent film.
  Control gel: Initially, the pressure ulcer was cleaned with saline. With the aid of a paper ruler, the ulcer was measured and photographed, as the ruler included the date and the initials of the patient. After measuring, a quantity of 5 grams of control gel was placed on the pressure ulcer and covered with sterile gauze and a transparent film.
  The curative was changed once a day during the treatment period, unless there was leakage of fluid, contamination, or signs of infection. Every three days the pressure ulcers of all patients were measured and photographed again, resulting in a total of six measurements per patient. The photos of pressure ulcers were evaluated for measurement of pressure ulcers and any kind of irritation.
Period: Overall Study
Arm/Group | Gel With HPβCD-I Complex | Gel With Insulin | Control Gel
Started | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gel With HPβCD-I Complex | Gel With Insulin | Control Gel | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Customized [Number; unit: participants]
  >45 and <75 years | 5 | 5 | 5 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 9
  Male | 2 | 3 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Index (%EI)
Description: Every three days the pressure ulcers (PUs) of all patients were measured and photographed again, resulting in a total of six measurements per patient. The photos were evaluated for measurement of PUs and any kind of irritation. At the end of this stage, the properly gathered study data was interpreted using the analysis software Mobile Wound Analyzer® (MOWA). Healing efficacy indices (% EI) were calculated as percentage reduction in the wound size at days 3, 6, 9, 12 and 15 from treatment beginning (d0). The % EI of the wound size was calculated by the following equation: %EI= ((Vsp.day-Vi)/Vi))x100. Vsp.day refers to the diameter (mm) values measured at day 3, 6, 9,12 and 15, while Vi refers to the baseline value measured before treatment (d0). The most representative result of treatment efficacy was observed on day 15, therefore it was used to calculate the % EI. For each group assessed, it was calculated the mean % EI of the five patients, resulting in a single value.
Time Frame: Measured every 3 days for 15 days
Population: Brazilian, bedridden, of both genders, aged between 45 and 75 years old and diabetic or not. Hyperglycemic volunteers and those with pressure ulcers other than grade II were excluded from the study. Grade II pressure ulcers were selected as they are a superficial lesion, with little tissue loss, and allow easy visualization of healing.
Measure: Mean (95% Confidence Interval); unit: percentage (%)
Arm/Group | Gel With HPβCD-I Complex | Gel With Insulin | Control Gel
Number analyzed (Participants) | 5 | 5 | 5
percentage (%) | 82.76 [78.25 to 86.15] | 43.66 [39.73 to 47.03] | 14.58 [12.53 to 16.25]

2. Secondary Outcome: Blood Glucose Tests in Order to Assess Whether the Gel With Hydroxypropyl-beta-cyclodextrin Complexed With Insulin (HPβCD-I) or With Insulin Could Cause an Increase in the Rate of Insulin in the Blood of Patients
Description: Dosages were provided four times daily (04h, 10h, 16h and 22h) to each patient during the 15-day study period, giving a total of 60 doses. To obtain these dosages, a drop of blood of patients was placed on a colorimetric strip and blood glucose was measured with the use of an Accu Check Active® glucose meter. The mean of 60 dosages was calculated for each patient at the end of 15 days. For each group assessed, it was calculated the mean of the measurements of the five patients, resulting in a single value.
Time Frame: Assessed daily at 04 h, 10 h, 16 h and 22 h for 15 days
Population: Brazilian, bedridden, of both genders, aged between 45 and 75 years old and diabetic or not. Hyperglycemic volunteers and those with pressure ulcers other than grade II were excluded from the study.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Gel With HPβCD-I Complex | Gel With Insulin | Control Gel
Number analyzed (Participants) | 5 | 5 | 5
mg/dL | 167.20 [153.92 to 208.90] | 168.88 [155.12 to 209.39] | 196.07 [103.00 to 325.00]

ADVERSE EVENTS:
Arm/Group | Gel With HPβCD-I Complex | Gel With Insulin | Control Gel
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Small numbers of subjects analyzed because of the type of pressure ulcer selected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No